CLINICAL TRIAL: NCT07069816
Title: Esophageal Motility and Gastric Emptying Disorders Among Different Thyroid Dysfunction
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa mohamed galal ahmed, GIT disorders among different thyroid dysfunction, Assiut University
Other Study IDs: GIT and thyroid dysfunction
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: GI Disorders
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Scintigraphy — non invasive method in which the test meals and acquisition procedures have been standardized and the results are largely operator independent
Radiation: Scintigraphy — Non invasive method in which the test meals and acquisition procedures have been standardized

SUMMARY:
Detect prevalence of different gastroparesis symptoms among different thyroid disorders Effect of thyroid disorders either hypothyroidism, hyperthyroidism and subclinical disorders in upper gastro motility

ELIGIBILITY:
Inclusion Criteria:

* all patient diagnosed as hypothyroidism, hyperthyroidism and subclinical thyroid disorders in diabetic and endocrinological centre in Assiut university hospitals, age above 18 years

Exclusion Criteria:

* patients take any drugs affect GIT motility Patients with acute infection Patients with major surgeries or recent trauma less than 6 months Patients known to have malignancy Patients with previous history of bariatric surgery Patients with history of liver cirrhosis or inflammatory bowel diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patient diagnosed as hypothyroidism, hyperthyroidism and subclinical thyroid disorders, age above 18 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Detect prevalence of different gastroparesis symptoms among different thyroid disorders | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Esraa, Asyut, Egypt